CLINICAL TRIAL: NCT02477215
Title: Phase I/II Study of Bendamustine and IXAZOMIB (MLN9708) Plus Dexamethasone in Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Bendamustine and IXAZOMIB (MLN9708) Plus Dexamethasone in Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Parameswaran Hari (Other)
Responsible Party: Sponsor-Investigator, Parameswaran Hari, Section Head, Hematological Malignancies Director, Adult Blood and Marrow Transplant Program, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00024991
Record Dates: First submitted 2015-06-12; First posted 2015-06-22 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Dexamethasone; Calcium Dobesilate; Bendamustine Hydrochloride; Maximum Tolerated Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MLN9708, Bendamustine and Dexamethasone Dose Escalation (Experimental): Ixazomib 4 mg, days 1, 8, 15.
  Dexamethasone 40 mg oral weekly.
  Bendamustine dose levels: 70 mg/m^2, 80mg/m^2, or 90 mg/m^2 given on days 1 and 2
  Interventions: Drug: MLN9708; Drug: Dexamethasone; Drug: Bendamustine (multiple dose levels)
- MLN9708, Bendamustine and Dexamethasone MTD (Experimental): Ixazomib 4 mg, days 1, 8, 15.
  Dexamethasone 40 mg oral weekly.
  Bendamustine dose levels: MTD given on days 1 and 2
  Interventions: Drug: MLN9708; Drug: Dexamethasone; Drug: Bendamustine (MTD)

INTERVENTIONS:
Drug: MLN9708 — 4 mg of MLN9708 delivered on days 1, 8 and 15 of a 28 day cycle.
  Other Names: Ixazomib
Drug: Dexamethasone — 40 mg oral on Days 1, 8, 15 of each 28 day cycle.
  Other Names: Decadron
Drug: Bendamustine (multiple dose levels) — 70 mg/m^2, 80 mg/m^2, or 90 mg/m^2 on days 1 and 2
  Other Names: Treanda; Treakisym; Ribomustin
  Arms: MLN9708, Bendamustine and Dexamethasone Dose Escalation
Drug: Bendamustine (MTD) — 80 mg/m^2 on days 1 and 2
  Other Names: Treanda; Treakisym; Ribomustin
  Arms: MLN9708, Bendamustine and Dexamethasone MTD

SUMMARY:
This Phase I/II study is designed to first identify doses of MLN9708 and bendamustine that are associated with an acceptable adverse event profile when delivered together in 28-day cycles. Additionally, the study aims to assess the efficacy of the combination in patients with relapsed/refractory multiple myeloma. Responders (stable disease or more), will continue to receive up to eight cycles total in the absence of further progressive disease.

DETAILED DESCRIPTION:
OVERVIEW: This Phase I/II study is designed to first identify doses of MLN9708 and bendamustine that are associated with an acceptable adverse event profile when delivered together in 28-day cycles. Additionally, the study aims to assess the efficacy of the combination in patients with relapsed/refractory multiple myeloma. Responders (stable disease or more),will continue to receive up to eight cycles total in the absence of further progressive disease.

OVERVIEW OF THE DOSE ESCALATION/DE-ESCALATION: This study aims to assess the combination's efficacy in patients with relapsed/refractory multiple myeloma. Responders (stable disease or more) will continue to receive up to eight cycles total in the absence of further progressive disease. The dose of MLN9708 will be fixed at 4 mg given on days 1, 8 and 15. Dexamethasone will be administered at 40 mg (oral) on Days 1, 8, 15 of each 28 day cycle. Dexamethasone administered as 40 mg oral on Days 1, 8, 15 of each 28 day cycle. Three doses of bendamustine will be evaluated (Dose 1: 70 mg/m^2, days 1 and 2; Dose 2: 80 mg/m^2. days 1 and 2; and Dose 3: 90 mg/m^2, days 1 and 2).

PHASE 1 DESIGN: A 3+3 design was employed. At each dose, three patients were initially evaluated. When no dose limiting toxicities were observed, the bendamustine dose will be increased.

PHASE 2 DESIGN: Design for Phase II portion of study: The MTD or a recommended phase 2 dose (RP2D) for the combination. The plan is to treat additional patients at that dose to assess efficacy and response to treatment. The investigators plan to enroll 19 patients (including those treated at the MTD in Phase I).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female patients 18 years or older.
2. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
3. Female patients who:

   * Are postmenopausal for at least one year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice two effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR • Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

   Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
4. Patients must have have histologically or cytologically confirmed symptomatic Multiple Myeloma, who are non-responsive to or ineligible for autologous stem cell transplant, and who progress after prior exposure to proteasome inhibitor (bortezomib, carfilzomib) and lenalidomide or pomalidomide or thalidomide (IMID); and refractory/progressing to at least one of these agents and must meet at least one of the following parameters of measurable disease:

   * Measurable levels of monoclonal protein (M protein): > 1 g/dL of immunoglobin G (IgG) or immunoglobin M (IgM) M-protein or > 0.5 g/dL immunoglobin A (IgA) or immunoglobin D (IgD) M protein on serum protein electrophoresis OR > 200 mg/24h of free light chain proteinuria on a 24 hour urine protein electrophoresis which must be obtained within 4 weeks prior to registration OR > 10 mg/dL involved free light chain on serum free light chain testing with an abnormal kappa:lambda light chain ratio.
   * Patients with lytic bone disease, defined as at least one lytic lesion that can be accurately measured in at least one dimension.
5. Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2.
6. Patients are eligible after autologous or allogeneic stem cell transplantation. Allogeneic transplantation can be enrolled only if they have no ongoing transplant related side effects.
7. Patients must be at least 2 weeks from major surgery, radiation therapy, participation in other investigational trials and have recovered from clinically significant toxicities of these prior treatments
8. Patients must meet the following clinical laboratory criteria:

   * Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3. Platelet transfusions or granulocyte-colony stimulating factor (G-CSF) can be used to help patients meet eligibility criteria but are not allowed within 3 days before study enrollment.
   * Total bilirubin < 1.5 x the upper limit of the normal range (ULN), , OR, direct bilirubin within normal limits (WNL), when total bilirubin is >>< 1.5 x the ULN.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x ULN.
   * Calculated creatinine clearance ≥ 30 mL/min.

EXCLUSION CRITERIA

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
2. Failure to have fully recovered (ie, ≤ Grade 1 toxicity) from the reversible effects of prior chemotherapy except for peripheral neuropathy, which is addressed in exclusion criteria no. #14.
3. Major surgery within 14 days before enrollment.
4. Radiotherapy within 14 days before enrollment. If the involved field is limited (single disease focus not involving pelvis and involving <36 Gy radiation), 7 days will be considered a sufficient interval between treatment and administration of Ixazomib provided hematologic inclusion parameters are met.
5. Central nervous system involvement.
6. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
7. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
8. Systemic treatment, within 14 days before the first dose of IXAZOMIB, with strong inhibitors of cytochrome P1A2 (CYP1A2) (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P3A (CYP3A) (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
9. Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
10. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
11. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
12. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of IXAZOMIB including difficulty swallowing.
13. Diagnosed or treated for another malignancy where the expected survival is less than two years will be excluded. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
14. Patient has ≥ Grade 2 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
15. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
16. Patients that have previously been treated with IXAZOMIB, or participated in a study with IXAZOMIB whether treated with IXAZOMIB or not.
17. Patients with a history of severe chronic obstructive pulmonary disease requiring ongoing oxygen support or those with a resting oxygen saturation <92% on room air irrespective of the cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2020-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Hari, MD, MRCP, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bendamustine (70 mg/m^2), MLN9708, Dexamethasone: MLN9708 : 4 mg, days 1, 8, 15.
  Dexamethasone: 40 mg oral weekly.
  Bendamustine: 70 mg/m^2 days 1 and 2
- Bendamustine (80 mg/m^2), MLN9708, Dexamethasone: MLN9708 : 4 mg, days 1, 8, 15.
  Dexamethasone: 40 mg oral weekly.
  Bendamustine: 80 mg/m^2 days 1 and 2
- Bendamustine (90 mg/m^2), MLN9708, Dexamethasone: MLN9708 : 4 mg, days 1, 8, 15.
  Dexamethasone: 40 mg oral weekly.
  Bendamustine: 90 mg/m^2 days 1 and 2
Period: Dose Escalation Phase
Arm/Group | Bendamustine (70 mg/m^2), MLN9708, Dexamethasone | Bendamustine (80 mg/m^2), MLN9708, Dexamethasone | Bendamustine (90 mg/m^2), MLN9708, Dexamethasone
Started | 4 | 8 | 6
Completed | 3 | 6 | 6
Not Completed | 1 | 2 | 0
Not completed — Physician Decision | 1 | 2 | 0
Period: Fixed Dose Phase
Arm/Group | Bendamustine (70 mg/m^2), MLN9708, Dexamethasone | Bendamustine (80 mg/m^2), MLN9708, Dexamethasone | Bendamustine (90 mg/m^2), MLN9708, Dexamethasone
Started | 0 (No subjects were started in this group as it was not the optimal dose.) | 20 (Subjects in Period 1 did not continue into Period 2. This is a new subject population.) | 0 (No subjects were started in this group as it was not the optimal dose.)
Completed | 0 | 13 | 0
Not Completed | 0 | 7 | 0
Not completed — Physician Decision | 0 | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation Phase: Bendamustine (70 mg/m^2), MLN9708, Dex.: MLN9708: 4 mg of MLN9708 delivered on days 1, 8 and 15 of a 28 day cycle.
  Dexamethasone: 40 mg oral on Days 1, 8, 15 of each 28 day cycle.
  Bendamustine: 70 mg/m^2 days 1 and 2
- Dose Escalation Phase: Bendamustine (80 mg/m^2), MLN9708, Dex.; Fixed Dose Phase: MLN9708: 4 mg of MLN9708 delivered on days 1, 8 and 15 of a 28 day cycle.
  Dexamethasone: 40 mg oral on Days 1, 8, 15 of each 28 day cycle.
  Bendamustine: 80 mg/m^2 days 1 and 2
- Dose Escalation Phase: Bendamustine (90 mg/m^2), MLN9708, Dex.: MLN9708: 4 mg of MLN9708 delivered on days 1, 8 and 15 of a 28 day cycle.
  Dexamethasone: 40 mg oral on Days 1, 8, 15 of each 28 day cycle.
  Bendamustine: 90 mg/m^2 days 1 and 2
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Phase: Bendamustine (70 mg/m^2), MLN9708, Dex. | Dose Escalation Phase: Bendamustine (80 mg/m^2), MLN9708, Dex. | Dose Escalation Phase: Bendamustine (90 mg/m^2), MLN9708, Dex. | Fixed Dose Phase | Total
Number analyzed (Participants) | 4 | 8 | 6 | 20 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 10 | 14
  >=65 years | 3 | 6 | 5 | 10 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 7 | 15
  Male | 2 | 6 | 2 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 8 | 6 | 19 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 7 | 8
  White | 4 | 7 | 5 | 13 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 8 | 6 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Bendamustine
Description: Maximum tolerated dose of bendamustine in combination with fixed doses of ixazomib (MLN9708) and dexamethasone will be determined from the incidence of dose limiting toxicities at each dosage.
Time Frame: Six months for each dosing cohort
Population: All participants received at least ne dose of Bendamustine at either 70 mg/m^2, 80 mg^2 or 90 mg/m^2.
Measure: Number; unit: mg/m^2
Groups:
- MLN9708, Bendamustine and Dexamethasone: MLN9708: 4 mg of MLN9708 delivered on days 1, 8 and 15 of a 28 day cycle.
  Dexamethasone: 40 mg oral on Days 1, 8, 15 of each 28 day cycle.
  Bendamustine:70 mg/m^2, 80 mg/m^2, or 90 mg/m^2 on days 1 and 2
Arm/Group | MLN9708, Bendamustine and Dexamethasone
Number analyzed (Participants) | 15
mg/m^2 | 80

2. Primary Outcome: Objective Response Rate
Description: Objective response rate was defined as the number of subjects achieving a complete response (CR) or partial response (PR) after at least four cycles of ixazomib (MLN9708) and bendamustine plus dexamethasone.
Time Frame: 18 months
Population: Subjects receiving the fixed dose of 80 mg/m^2 Bendamustine were included in this analysis. Results from five of the subjects in the Dose Escalation Phase of this study who also received 80 mg/m^2 Bendamustine were included in the analysis. One of the Dose Expansion Phase subjects did not complete sufficient dosing cycles for inclusion.
Measure: Number; unit: participants
Groups:
- MLN9708, Bendamustine and Dexamethasone: Ixazomib 4 mg, days 1, 8, 15.
  Dexamethasone 40 mg oral weekly.
  Bendamustine dose levels: 80mg/m2 days 1,2
  MLN9708: 4 mg of MLN9708 delivered on days 1, 8 and 15 of a 28 day cycle.
  Dexamethasone: 40 mg oral on Days 1, 8, 15 of each 28 day cycle.
  Bendamustine: 80mg/m2 days 1,2
Arm/Group | MLN9708, Bendamustine and Dexamethasone
Number analyzed (Participants) | 18
participants | 11

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was determined as the average number of months subjects survived following enrollment.
Time Frame: 36 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: MONTHS
Groups:
- MLN9708, Bendamustine and Dexamethasone: MLN9708: 4 mg of MLN9708 delivered on days 1, 8 and 15 of a 28 day cycle.
  Dexamethasone: 40 mg oral on Days 1, 8, 15 of each 28 day cycle.
  Bendamustine: 80 mg/m^2 days 1,2
Arm/Group | MLN9708, Bendamustine and Dexamethasone
Number analyzed (Participants) | 18
MONTHS | 23.2 [16.3 to 30.07]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: This measure is the number of months participants remain free from evidence of disease.
Time Frame: 18 months
Population: For this analysis, all 20 participants who received the fixed dose of 80 mg/m^2 Bendamustine and all 8 participants who received Bendamustine (80 mg/m^2) in the Dose Escalation phase, were combined.
Measure: Median (95% Confidence Interval); unit: MONTHS
Arm/Group | MLN9708, Bendamustine and Dexamethasone
Number analyzed (Participants) | 28
MONTHS | 5.2 [1.96 to 8.3]

5. Secondary Outcome: Cumulative Response Rates in Patients After Eight Cycles.
Description: Percentage of subject response rates at any point during the eight cycles.
Time Frame: 18 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | MLN9708, Bendamustine and Dexamethasone
Number analyzed (Participants) | 18
percentage of participants | 28

6. Secondary Outcome: Duration of Response (DoR)
Description: Median time in months participants maintain CR, PR or stable disease.
Time Frame: 36 months
Population: as for outcome 2
Measure: Median (Full Range); unit: MONTHS
Arm/Group | MLN9708, Bendamustine and Dexamethasone
Number analyzed (Participants) | 18
MONTHS | 5.1 [1 to 5.2]

7. Secondary Outcome: Number of Participants Experiencing Dose-Limiting Toxicity (DLT)
Description: A 3+3 design was employed. At each dose, three patients were initially evaluated. If no dose limiting toxicities were observed, the bendamustine dose was increased; if one dose limiting toxicity is observed, three additional patients were treated at that dose. A dose at which 2 DLTs were observed in 3 or 6 patients were judged to be too toxic and the lower dose was defined as the maximally tolerated dose (MTD).
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine (70 mg/m^2), MLN9708, Dexamethasone | Bendamustine (80 mg/m^2), MLN9708, Dexamethasone | Bendamustine (90 mg/m^2), MLN9708, Dexamethasone
Number analyzed (Participants) | 3 | 6 | 6
Participants | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Bendamustine (70 mg/m^2), MLN9708 and Dexamethasone: MLN9708: 4 mg of MLN9708 delivered on days 1, 8 and 15 of a 28 day cycle.
  Dexamethasone: 40 mg oral on Days 1, 8, 15 of each 28 day cycle.
  Bendamustine: 70 mg/m^2 on days 1 and 2
- Bendamustine (80 mg/m^2), MLN9708 and Dexamethasone: MLN9708: 4 mg of MLN9708 delivered on days 1, 8 and 15 of a 28 day cycle.
  Dexamethasone: 40 mg oral on Days 1, 8, 15 of each 28 day cycle.
  Bendamustine: 80 mg/m^2 on days 1 and 2.
  This reporting group includes subjects from both the Dose Escalation and Fixed Dose Phases who received Bendamustine at 80 mg/m^2.
- Bendamustine (90 mg/m^2), MLN9708 and Dexamethasone: MLN9708: 4 mg of MLN9708 delivered on days 1, 8 and 15 of a 28 day cycle.
  Dexamethasone: 40 mg oral on Days 1, 8, 15 of each 28 day cycle.
  Bendamustine: 90 mg/m^2 on days 1 and 2
Arm/Group | Bendamustine (70 mg/m^2), MLN9708 and Dexamethasone | Bendamustine (80 mg/m^2), MLN9708 and Dexamethasone | Bendamustine (90 mg/m^2), MLN9708 and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 2/3 | 8/19 | 2/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 8/19 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 0/19 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (70 mg/m^2), MLN9708 and Dexamethasone (N=3) | Bendamustine (80 mg/m^2), MLN9708 and Dexamethasone (N=19) | Bendamustine (90 mg/m^2), MLN9708 and Dexamethasone (N=6)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Mobitz type 1 (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Exacerbated COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT02477215/Prot_SAP_000.pdf